CLINICAL TRIAL: NCT02711826
Title: Treg Adoptive Therapy in Subclinical Inflammation in Kidney Transplantation (CTOT-21)
Brief Title: Treg Therapy in Subclinical Inflammation in Kidney Transplantation
Acronym: TASK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-21
Record Dates: First submitted 2016-03-11; First posted 2016-03-17 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Adult Living Donor Kidney Transplant Recipients; Renal Transplant; Living Kidney Donor
Keywords: graft inflammation; Treg; polyclonally expanded Tregs (polyTregs); calcineurin inhibitors (CNIs); mTOR inhibitors
MeSH Terms: interventions — Everolimus; Tacrolimus; Mycophenolic Acid; Acetaminophen; Diphenhydramine; Biopsy; Blood Specimen Collection; Phlebotomy; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance CNI based immunosuppression therapy group (Active Comparator): Standard of care
  (N=7 participants in this group)
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Mycophenolic acid; Procedure: Biopsy, Kidney; Procedure: Blood Draw
- Polyclonal Regulatory T Cells group (Experimental): Subjects to receive polyTregs (550 ± 450 x 10^6). After receiving at least 300X10^6 polyTregs infusion, eligible subjects will start mammalian Target of Rapamycin (mTOR) inhibitor.
  Target tacrolimus trough levels prior to conversion to everolimus are 4-11 μg/dl, which falls within standard of care. For eligible participants in polyTregs and darTregs groups, the tacrolimus dose will be reduced by 50% when everolimus is initiated. Tacrolimus will be discontinued 4 weeks after initiation of everolimus therapy.
  Everolimus, a mTOR inhibitor immunosuppressant, will be initiated at a dose of 1.5 mg orally twice daily and titrated, as needed. Participants will begin everolimus with target trough levels of 3-8μg/L for 4 weeks while still taking tacrolimus. Everolimus target trough levels will be 6-10 μg/L when tacrolimus is discontinued.
  (N=7 participants in this group)
  Interventions: Biological: Polyclonal Regulatory T Cells; Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Mycophenolic acid; Drug: Acetaminophen; Drug: Diphenhydramine; Procedure: Biopsy, Kidney; Procedure: Blood Draw; Procedure: Leukapheresis; Procedure: IS regimen conversion

INTERVENTIONS:
Biological: Polyclonal Regulatory T Cells — Participants randomized to polyTregs group will receive a single infusion of 550 ± 450 x 10^6 polyTregs.
  Other Names: Polyclonal Tregs; polyTregs
  Arms: Polyclonal Regulatory T Cells group
Drug: Everolimus
  Other Names: Zortress
  Arms: Polyclonal Regulatory T Cells group
Drug: Tacrolimus
  Other Names: FK-506; FR-900506; Prograf
Drug: Mycophenolate mofetil — All enrolled participants will be on MMF (or MPA below) at the time of study entry at a minimum dose of 1000mg per day.
  Other Names: Cellcept; MMF
Drug: Mycophenolic acid — All enrolled participants will be on MPA (or MMF above) at the time of study entry at a minimum dose of 720mg per day.
  Other Names: Myfortic; MPA
Drug: Acetaminophen — 650 mg acetaminophen, administered 30-60 minutes prior to infusion as pre-medication.
  Other Names: Tylenol
  Arms: Polyclonal Regulatory T Cells group
Drug: Diphenhydramine — 25-50 mg diphenhydramine intravenously or by mouth, administered 30-60 minutes prior to infusion as pre-medication.
  Other Names: Benadryl
  Arms: Polyclonal Regulatory T Cells group
Procedure: Biopsy, Kidney
  Other Names: Kidney Biopsy
Procedure: Blood Draw
  Other Names: Phlebotomy; Venipuncture
Procedure: Leukapheresis
  Other Names: leukocytapheresis
  Arms: Polyclonal Regulatory T Cells group
Procedure: IS regimen conversion — Conversion from Tacrolimus, a calcineurin inhibitors (CNI), to Everolimus, an mTOR inhibitor.
  Other Names: Everolimus Conversion
  Arms: Polyclonal Regulatory T Cells group

SUMMARY:
The purpose of this study is:

* To see if polyTregs can reduce inflammation in a transplanted kidney.
* To find out what effects, good or bad, polyTregs will have in the kidney recipient.
* To find out what effects, good or bad, taking everolimus after polyTregs will have in the kidney recipient.

DETAILED DESCRIPTION:
Inflammation occurs when the body's defense system recognizes a foreign object (such as a transplanted kidney), and responds by sending white blood cells to attack the foreign object. These cells and the substances they produce can damage the transplanted kidney. There is currently no standard treatment for inflammation in the kidney; some transplant centers do not treat inflammation at all. Rejection is a more severe form of inflammation and injury. Both inflammation and rejection are diagnosed by looking at a piece of kidney (a kidney biopsy) under a microscope. Kidneys that have inflammation and/or rejection do not work as well or last as long as kidneys without injury.

People who have a transplant take immunosuppressive drugs (IS) to prevent inflammation and rejection. Although kidney transplant recipients usually do well in the first five years after transplant, transplant researchers are interested in finding ways to prevent inflammation and rejection without IS, or with lower doses of IS in order to avoid side effects.

While some white blood cells cause inflammation, other types of white blood cells, called T regulatory cells (Tregs), can control inflammation. Tregs may have an important role in controlling or preventing inflammation and rejection. A person's Tregs can be grown in the laboratory to increase their number (polyTreg). These Tregs can be given back through a needle placed in a vein (IV). PolyTregs, when given to the recipient, might reduce inflammation in the transplanted kidney. However, this effect has not yet been shown.

One of the IS drugs used in kidney transplant is Everolimus. Everolimus has been shown to help Tregs survive better than other types of IS drugs.

This is a randomized open-label trial to determine the safety and efficacy of a single dose of autologous polyTregs in renal transplant recipients with subclinical inflammation (SCI) in the 3 to 7 months post-transplant allograft protocol biopsy compared to control patients treated with CNI-based immunosuppression. The efficacy of the Treg therapy will be assessed by the reduction of graft inflammation on biopsies performed at 7 months after study group allocation compared to the eligibility biopsy.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Subject must be able to understand and provide informed consent;
2. Age ≥18 years of age at the time of study entry;
3. Recipients of non- Human Leukocyte Antigen (HLA) identical living or deceased renal transplants;
4. Protocol renal allograft biopsy at 5 months (± 8 weeks) after transplantation with Banff i1 and/or ti1 with concomitant t scores t0, t1,t2 or t3; Banff i2 and/or ti2 with concomitant t scores t0 or t1; and without v > 0, [ptc + g] ≥2, C4d >1 (by immunofluorescence, IF), or C4d > 0 (by immunohistochemistry, IHC); confirmed by central pathologist. Subjects must not be treated for pathologic criteria (e.g. steroids).
5. Estimated glomerular filtration rate (eGFR) ≥30 ml/min at the time of study entry;
6. Maintenance immunosuppression consisting of tacrolimus, MMF/MPA (≥1000 mg/720 mg daily) ± prednisone (≤10 mg/day);
7. Current immunizations including TdAP, hepatitis B, pneumococcal and seasonal influenza vaccines prior to study treatment, completed prior to randomization and no less than 14 days prior to planned manufacturing collection;
8. Documented Hepatitis B (HB) serologies must be:

   1. Positive HB surface antibody, negative HB core antibody and negative HB surface antigen for recipients immune to hepatitis B
   2. Negative HB surface antibody, negative HB core antibody and negative HB surface antigen for non-immune/ HBV naïve recipients provided donor had negative HB core antibody and negative HB surface antigen at the time of donation.
9. Negative TB test (PPD, interferon-gamma release assay, ELISPOT testing) within 1 year prior to enrollment. Subjects with a history of TB (positive TB test without active infection) must have completed one of the latent TB infection treatment regimens endorsed by the CDC (Division of TB Elimination, 2016). Alternative regimens for latent TB infection eradication will be adjudicated by the site's infectious disease specialist.
10. Female subjects of childbearing potential must have reviewed the Mycophenolate Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) and have a negative pregnancy test upon study entry (Reference:https://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafetyInformationforPatientsandProviders/ucm318880.htm); and
11. Female subjects with child-bearing potential, must agree to use FDA approved methods of birth control for the duration of the study; subjects must consult with their physician and determine the most suitable method(s) that are greater than 80% effective (http://www.fda.gov/birthcontrol).

Treg Infusion Inclusion Criteria:

1. Individuals randomized to the polyTreg and darTreg groups who continue to meet all of the enrollment criteria; and
2. Negative SARS-COV2 by RTP-PCR testing within 1 week of Treg infusion.

mTOR Conversion Inclusion Criteria:

Individuals who meet all of these criteria are eligible for mTOR conversion:

1. Received at least 300 x 10^6 polyTreg infusion;
2. Resolution of inflammation on the 2 week post-infusion biopsy as compared to the baseline biopsy, confirmed by central pathologist.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
2. History of malignancy; except adequately treated basal cell carcinoma;
3. History of graft loss from acute rejection within 1 year after any previous transplant;
4. History of transplant renal artery stenosis;
5. History of cellular rejection prior to enrollment that did not respond to steroids and/or subsequent creatinine after treatment for rejection greater than 15% above baseline;
6. Known hypersensitivity to mTOR inhibitors or contraindication to everolimus (including history of wound healing complications);
7. Any chronic illness requiring uninterrupted anti-coagulation after kidney transplantation;
8. Post-transplant DSA >5000 MFI or post-transplant treatment with IVIg for DSA.

   * Note: Enrolled subjects with post-transplant DSA >2000 MFI will not be eligible for mTOR conversion.
9. Positive HIV 1 or HIV 2 serology prior to transplantation;
10. Positive HBSAg or HBcAb serology;
11. Proteinuria with urine protein-to-creatinine ratio > 1.0 g/g;
12. Any condition requiring chronic use of corticosteroids >10mg/day at the time of study entry;
13. Subjects requiring treatment for pathologic findings on study eligibility biopsy (see inclusion 5).
14. Active infection at the time of study entry;
15. History of active TB or latent TB without adequate treatment;
16. Serum BK virus >1,000 copies/ml by Polymerase Chain Reaction (PCR) at the time of study entry;
17. Hematocrit <27%; Absolute Neutrophil Count (ANC) < 1,000/μL; and/or lymphocyte count <500/μL at the time of study entry;
18. Participation in any other studies with investigational drugs or regimens in the preceding year;
19. Any condition or prior treatment which, in the opinion of the investigator, precludes study participation.
20. Unable to provide adequate biopsy specimen (paraffin embedded formalin fixed) from eligibility biopsy (3-7 months post -transplant) for quantitative analysis.
21. Epstein-Barr virus (EBV) naïve recipient of a kidney from an EBV positive donor; and/or historically EBV naïve recipient with primary EBV infection at the time of screening (e.g., anti-VCA IgM positive and EBNA negative), a positive EBV PCR.
22. Hepatitis C Virus AB positive subjects with negative HCV PCR are eligible if they have spontaneously cleared infection or are in sustained virologic remission for at least 12 weeks after treatment.
23. Positive SARS-CoV2 testing by RT-PCR

Treg Infusion Exclusion Criteria:

Individuals randomized to polyTreg and darTreg groups who meet any of these criteria are not eligible for Treg infusion:

1. Received any vaccination within 14 days prior to blood collection for Treg manufacture;
2. Unacceptable Treg product;
3. Positive pregnancy test for women of child bearing potential.

mTOR Conversion Exclusion Criteria:

1. Post-transplant Donor-Specific Antibodies (DSA) >2000 mean florescence intensity (MFI).
2. Any condition or clinical variable, which in the opinion of the site investigator, precludes conversion to mTOR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, MD, Principal Investigator — University of California at San Francisco; Sindhu Chandran, MD, Study Chair — University of California at San Francisco
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - University of Colorado Health Transplant Center - Anschutz, Aurora, Colorado
  - Northwestern University Comprehensive Transplant Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort [https://immport.niaid.nih.gov/ ], a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts, upon completion of the study.

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 adult, kidney transplant candidates were enrolled across 7 US sites between September 2016 and May 2022. Of these 27 enrolled transplant candidates, 18 participants were randomized and 16 initiated study treatment. Additionally, 5 living donors consented at 2 US sites between September 2016 and September 2018.
Pre-assignment Details: Potential participants signed informed consent before undergoing any study procedures. Screening criteria, including results from a 5 month post-transplant standard of care biopsy, were evaluated to determine study eligibility and candidacy for randomization. Living donors were asked to consent for a blood draw and minimal medical information.
Groups:
- Maintenance: Participants in this group continued standard CNI-based maintenance immunosuppression therapy with no intervention.
- polyTregs: Participants in the polyclonally expanded regulatory T cells (polyTregs) group received a single infusion of 550 ± 450 x 10⁶ polyTregs administered via a peripheral intravenous line primed with saline by gravity in approximately 20 to 30 minutes.
- darTregs: Participants in the donor alloantigen reactive regulatory T cells (darTregs) group received a single infusion of 400 ± 100 x 10⁶ darTregs administered via a peripheral intravenous line primed with saline by gravity in approximately 20 to 30 minutes.
- Enrolled, Discontinued Pre-Randomization: Participants who failed screening or were eligible but did not proceed to randomization.
- Enrolled, Living Donor: Living donors of the prospective transplant recipient were consented and enrolled into the study.
Period: Overall Study
Arm/Group | Maintenance | polyTregs | darTregs | Enrolled, Discontinued Pre-Randomization | Enrolled, Living Donor
Started | 3 | 9 (Neither of the two not completed participants received infusion of the cellular product; one was reassigned to the Maintenance group because of no longer meeting infusion criteria due to active infection.) | 6 (None of the five not completed participants received infusion of the cellular product; 4 were reassigned to the Maintenance group because of failure to manufacture the cellular product.) | 9 | 5
Completed | 3 | 7 | 1 | 0 | 5
Not Completed | 0 | 2 | 5 | 9 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 4 | 0
Not completed — Failure to manufacture cellular product | 0 | 0 | 5 | 0 | 0
Not completed — Infusion canceled for active infection | 0 | 1 | 0 | 0 | 0
Not completed — Screen failures | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population who initiated study treatment, reflecting reassignment of participants from either the polyTregs or darTregs group to the Maintenance group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maintenance | polyTregs | darTregs | Enrolled, Living Donor | Total
Number analyzed (Participants) | 8 | 7 | 1 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 1 | 4 | 18
  >=65 years | 1 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (11.78) | 52.1 (11.94) | 58.0 (0.00) | 48.0 (17.66) | 49.7 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 0 | 3 | 11
  Male | 4 | 3 | 1 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 1 | 6
  Not Hispanic or Latino | 6 | 4 | 1 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 1 | 4
  White | 5 | 2 | 1 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 0 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 1 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Banff 2A or Higher Acute Cell-mediated Rejection and/or Acute Antibody Mediated Rejection
Description: Acute cell-mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 2A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2A, 2B, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection. Antibody mediated rejection was defined as diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury.
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated study treatment, subset to participants with available central pathology read data.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 6 | 7 | 1
Participants | 0 | 0 | 0

2. Primary Outcome: Timing of Banff 2A or Higher Acute Cell-mediated Rejection and/or Acute Antibody Mediated Rejection
Description: Acute cell-mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 2A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2IA, 2IB, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection. Antibody mediated rejection was defined as diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury.
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated study treatment, subset to participants with available central pathology read data who had severe acute cell-mediated rejection and/or acute antibody mediated rejection. No participants met the criteria for inclusion in this analysis population.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Incidence of Study Defined Grade 3 or Higher Infection
Description: This outcome measure includes infections reported as adverse events. Severe infection was defined in the study as a Grade 3 or higher infection. Severity is graded as 1 through 5, with 1 being least severe to 5 being most severe. Grade 3 is any infection associated with hemodynamic compromise requiring pressors; any infection necessitating ICU level of care; any infection necessitating operative intervention; any infection involving the central nervous system; any infection with a positive fungal blood culture; any proven or probable aspergillus infection; any tissue invasive fungal infection; any pneumocystis jiroveci infection. Grade 4 is any life-threatening infection. Grade 5 is any infection resulting in death.
Time Frame: 405 days after randomization for participants in the maintenance group; 365 days after Treg infusion for the participants in the polyTregs or darTregs groups
Population: Intent-to-treat population who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 8 | 7 | 1
Participants | 2 | 3 | 1
Statistical Analysis 1: Comparison: Maintenance vs polyTregs vs darTregs; Test type: Superiority; p = 0.425, Fisher Exact

4. Primary Outcome: Timing of Study Defined Grade 3 or Higher Infection
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Intent-to-treat population who initiated study treatment and experienced a severe infection
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 2 | 3 | 1
Days | 179.0 [99.0 to 259.0] | 116.0 [36.0 to 179.0] | 84.0 [84.0 to 84.0]
Statistical Analysis 1: Comparison: Maintenance vs polyTregs vs darTregs; Test type: Superiority; p = 0.700, Kruskal-Wallis

5. Primary Outcome: Percent Change in Inflammation
Description: The change in inflammation was measured by the percentage area of the renal cortex occupied by inflammatory cells on biopsy 7 months after group allocation. This change was expressed as the percent change relative to the baseline biopsy. The measurements were obtained using computer-assisted quantitative image analysis.
Time Frame: At baseline biopsy and at 7 months post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants from the Maintenance and polyTregs groups with available LCA data from the biopsy 7 months post-group allocation. darTregs group excluded from efficacy analysis per the protocol and statistical analysis plan.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 4 | 6 | 0
Percent change | -59.16 [-70.65 to -35.35] | -78.95 [-85.41 to -68.11] |
Statistical Analysis 1: Comparison: Maintenance vs polyTregs; Test type: Superiority; p = 0.201, Kruskal-Wallis

6. Primary Outcome: Immunologic Profiles of Kidney Transplant Recipients
Description: CRM (Common Response Module) score is a geometric mean of CRM gene expression. This score is used to identify evidence of rejection or inflammation in participants at the time of biopsy.
Time Frame: At 2 weeks post-polyTregs infusion (for polyTregs infusion group) and at 7 months post-group allocation (both groups)
Population: Data were not collected for this endpoint.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Incidence of polyTregs Infusion Reactions
Description: An infusion reaction is characterized by an adverse reaction to the infusion of pharmacological substance, as defined using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 set forth by the National Cancer Institute.
Time Frame: 365 days after Treg infusion for the participants in the polyTregs group
Population: Intent-to-treat population, subset to participants who received the polyTregs infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 7 | 0
Participants |  | 0 |

8. Secondary Outcome: Severity of polyTregs Infusion Reactions
Description: Severity of infusion reactions were defined using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 set forth by the National Cancer Institute. Severity of adverse events is graded as 1 through 5, with 1 being least severe to 5 being most severe.
Time Frame: 365 days after Treg infusion for the participants in the polyTregs group
Population: Intent-to-treat population, subset to participants who received the polyTregs infusion and had a polyTregs infusion reaction. No participants met the criteria for inclusion in this analysis population.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Timing of polyTregs Infusion Reactions
Description: as for outcome 7
Time Frame: 365 days after Treg infusion for the participants in the polyTregs group
Population: as for outcome 8
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Incidence of Culture-proven and Clinically Diagnosed Infection.
Description: A culture-proven and clinically diagnosed infection in this study was defined as any locally reported infection due to bacterial organism, due to fungal organism, due to CMV, or which met adverse event criteria, except for COVID-19.
Time Frame: as for outcome 3
Population: Intent-to-treat population who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 8 | 7 | 1
Participants | 2 | 3 | 1

11. Secondary Outcome: Severity of Culture-proven and Clinically Diagnosed Infection
Description: A culture-proven and clinically diagnosed infection was defined as any locally reported infection due to bacterial organism, fungal organism, CMV, or which met adverse event criteria, except for COVID-19. Severe infection was defined in the study as a Grade 3 or higher infection. Severity is graded as 1 through 5 with 1 being least severe to 5 being most severe. Grade 3 is any infection associated with hemodynamic compromise requiring pressors; any infection necessitating ICU level of care; any infection necessitating operative intervention; any infection involving the central nervous system; any infection with a positive fungal blood culture; any proven or probable aspergillus infection; any tissue invasive fungal infection; any pneumocystis jiroveci infection. Grade 4 is any life-threatening infection. Grade 5 is any infection resulting in death. If a culture proven and clinically diagnosed infection did not qualify for AE reporting, then it did not have a severity grade.
Time Frame: as for outcome 3
Population: Intent-to-treat population who initiated study treatment, subset to those with culture-proven and clinically diagnosed infections
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 2 | 3 | 1
Participants
  Grade 3 | 2 | 2 | 1
  No Grade | 0 | 1 | 0

12. Secondary Outcome: Timing of Culture-proven and Clinically Diagnosed Infection
Description: A culture-proven and clinically diagnosed infection in this study was defined as any locally reported infection due to bacterial organism, fungal organism, CMV, or which met adverse event criteria, except for COVID-19.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 2 | 3 | 1
Days | 179.0 [99.0 to 259.0] | 179.0 [36.0 to 215.0] | 84.0 [84.0 to 84.0]

13. Secondary Outcome: Incidence of Acute Rejection Using Banff Grading
Description: Acute cell-mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 1A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2A, 2B, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection.
Time Frame: 405 days post-group allocation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 6 | 7 | 1
Participants | 0 | 0 | 0

14. Secondary Outcome: Severity of Acute Rejection Using Banff Grading
Description: as for outcome 13
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated study treatment, subset to participants with available central pathology read data and who experienced acute rejection. No participants met the criteria for inclusion in this analysis population.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Timing of Acute Rejection Using Banff Grading
Description: as for outcome 13
Time Frame: 405 days post-group allocation
Population: as for outcome 14
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Incidence of BK Viremia
Description: BK viremia was determined using locally reported serum PCR results. PCR results reported as positive and >0 copies/mL were considered as meeting the endpoint. Only positive results following Treg infusion were considered for participants in the polyTregs and darTregs groups.
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 8 | 7 | 1
Participants | 0 | 1 | 0

17. Secondary Outcome: Timing of BK Viremia
Description: as for outcome 16
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants who experienced BK viremia.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 1 | 0
Days |  | 365.00 [365.00 to 365.00] |

18. Secondary Outcome: Incidence of Cytomegalovirus (CMV) Reactivation
Description: CMV reactivation was defined as CMV viremia and determined using locally reported serum, plasma, or whole blood PCR results. PCR results reported as >0 IU/mL were considered as meeting the endpoint. Only positive results following Treg infusion were considered for participants in the polyTregs and darTregs groups.
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 8 | 7 | 1
Participants | 0 | 0 | 1

19. Secondary Outcome: Timing of CMV Reactivation
Description: as for outcome 18
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants who experienced CMV reactivation.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 1
Days |  |  | 84.0 [84.0 to 84.0]

20. Secondary Outcome: Incidence of > 10% Decrease in Estimated Glomerular Filtration Rate (eGFR) Compared to Baseline
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. eGFR was estimated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) 2021 equation. A value of 90+ means kidney function is normal. A value between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Values between 30 and 59 indicate moderately reduced kidney function. Values between 15 and 29 indicate severely reduced kidney function. Values below 15 indicate very severe or end stage kidney failure. The percent change in eGFR was calculated at each post-baseline timepoint as [(post-baseline eGFR minus baseline (i.e., screening) eGFR) divided by baseline eGFR] multiplied by 100 and rounded to the nearest hundredth for each participant. A participant was considered to have met the endpoint if at least one instance of a greater than 10% decrease from baseline was observed.
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 8 | 7 | 1
Participants | 5 | 6 | 1

21. Secondary Outcome: Timing of > 10% Decrease in eGFR Compared to Baseline
Description: as for outcome 20
Time Frame: 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants who had a >10% decrease in eGFR.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 5 | 6 | 1
Days | 51.0 [37.0 to 60.0] | 53.0 [30.0 to 64.0] | 44.0 [44.0 to 44.0]

22. Secondary Outcome: Incidence of Acute Rejection After Converting to mTOR Therapy Following polyTregs Infusion
Description: Acute cell-mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 2A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2A, 2B, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection.
Time Frame: 69 days post-group allocation to 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants who received the polyTregs infusion and converted to mTOR therapy. No participants met the criteria for inclusion in this analysis population.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Timing of Acute Rejection After Converting to mTOR Therapy Following polyTregs Infusion
Description: as for outcome 22
Time Frame: 69 days post-group allocation to 405 days post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants who received the polyTregs infusion, converted to mTOR therapy, and had an acute rejection event. No participants met the criteria for inclusion in this analysis population.
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Proportion of Participants Exhibiting >=25% Relative Decrease of Inflammation Between Baseline Kidney Biopsy and the Week 2 Kidney Biopsy
Description: The change in inflammation was measured by the percentage area of the renal cortex occupied by inflammatory cells on biopsy 2 weeks after polyTregs infusion. This change was expressed as the percent change relative to the baseline biopsy. The measurements were obtained using computer-assisted quantitative image analysis.
Time Frame: Baseline biopsy to week 2 kidney biopsy
Population: Intent-to-treat population who initiated treatment, subset to participants with available LCA data from the Week 2 biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 6 | 1
Participants | 0 | 2 | 0

25. Secondary Outcome: Proportion of Participants Exhibiting >=50% Relative Decrease of Inflammation Between Baseline Kidney Biopsy and the Week 2 Kidney Biopsy
Description: as for outcome 24
Time Frame: Baseline biopsy to week 2 kidney biopsy
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 0 | 6 | 1
Participants | 0 | 1 | 0

26. Secondary Outcome: Proportion of Participants Exhibiting >=25% Relative Decrease of Inflammation Between Baseline Kidney Biopsy and the 6 Month Kidney Biopsy
Description: The change in inflammation was measured by the percentage area of the renal cortex occupied by inflammatory cells on biopsy 7 months after study group allocation. This change was expressed as the percent change relative to the baseline biopsy. The measurements were obtained using computer-assisted quantitative image analysis.
Time Frame: Baseline biopsy to 7 months post-group allocation
Population: Intent-to-treat population who initiated treatment, subset to participants with available LCA data from the biopsy 7 months post-group allocation
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance | polyTregs | darTregs
Number analyzed (Participants) | 4 | 6 | 1
Participants | 3 | 5 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first study mandated procedure until a subject completes study participation (405 days after randomization for participants in the maintenance group; 365 days after treg infusion for the participants in the polyTregs or darTregs groups) or until 30 days after they prematurely withdraw (without withdrawing consent) or is withdrawn from the study.
Groups:
- polyTregs: Participants in the polyclonally expanded regulatory T cells (polyTregs) group received a single infusion of 550 ▒ 450 x 106 polyTregs administered via a peripheral intravenous line primed with saline by gravity in approximately 20 to 30 minutes.
- darTregs: Participants in the donor alloantigen reactive regulatory T cells (darTregs) group received a single infusion of 400 ▒ 100 x 106 darTregs administered via a peripheral intravenous line primed with saline by gravity in approximately 20 to 30 minutes.
Arm/Group | Maintenance | polyTregs | darTregs | Enrolled, Living Donor
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/8 | 4/8 | 1/2 | 0/5
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 0/2 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance (N=8) | polyTregs (N=8) | darTregs (N=2) | Enrolled, Living Donor (N=5)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance (N=8) | polyTregs (N=8) | darTregs (N=2) | Enrolled, Living Donor (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02711826/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02711826/SAP_003.pdf
  • Informed Consent Form: Donor ICF (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02711826/ICF_000.pdf
  • Informed Consent Form: Recipient ICF (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02711826/ICF_001.pdf